CLINICAL TRIAL: NCT03544749
Title: A Randomized Comparison of Ambu® AuraGain™ Laryngeal Mask Airway and I-gel in Patients With Simulated Cervical Immobilization
Brief Title: A Comparison of Ambu® AuraGain™ Laryngeal Mask Airway and I-gel in Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Clinical professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1803-124-932
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Laryngeal Mask; Intubation; Difficult or Failed

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambu® AuraGain™ group (Experimental)
  Interventions: Device: Ambu® AuraGain™
- I-gel group (Active Comparator)
  Interventions: Device: I-gel

INTERVENTIONS:
Device: Ambu® AuraGain™ — After induction of anesthesia, Ambu® AuraGain™ will be inserted for the mechanical ventilation.
  Arms: Ambu® AuraGain™ group
Device: I-gel — After induction of anesthesia, I-gel will be inserted for the mechanical ventilation.
  Arms: I-gel group

SUMMARY:
The supraglottic airway device(SAD), as an alternative to the endotracheal tube is inserted into the oral cavity and seals the upper esophagus and the surrounding tissue, effectively securing airway. SAD has evolved in recent years to increase efficiency and secure safety. The recently developed Ambu® AuraGain™ is a second-generation SAD with a built-in gastric port and is designed to be fitted well in the larynx and oral cavity after insertion because the shaft is bent at an angle of 90 degrees and has an inflatable cuff.

In a previous study, Ambu® AuraGain™ showed a higher sealing pressure and better fibreoptic finding compared to LMA Supreme in laparoscopic surgery.

On the other hand, I-gel and Ambu® AuraGain™, both of the second-generation SAD, show comparatively excellent performance according to the results of previous studies. However, there are no studies comparing the characteristics of two airway devices in adults.

The purpose of this study is to compare the performance of I-gel and Ambu® AuraGain™ to make a difficult airway-like situation using cervical collar for adult patients receiving mechanical ventilation under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing surgery under general anesthesia where supraglottic airway management will be appropriate.

Exclusion Criteria:

* Body mass index > 35 kg/m2
* High risk of regurgitation (hiatus hernia, gastro-esophageal reflux disease, non-fasting status)
* Criteria for difficult airway
* Patients with cervical disease or previous cervical spine surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | At an average of 30 seconds after insertion of laryngeal mask airway
  Oropharyngeal leak pressure is measured by closing the expiratory valve and administering fresh gas flow of 6 L/min, until the equilibrium pressure is reached (to a maximum of 40 cm of H2O).

SECONDARY OUTCOMES:
Oropharyngeal leak pressure | At 5 minute after insertion of laryngeal mask airway
  Oropharyngeal leak pressure is measured by closing the expiratory valve and administering fresh gas flow of 6 L/min, until the equilibrium pressure is reached (to a maximum of 40 cm of H2O).
The time for successful insertion of the device | During induction of anesthesia, an average of 60 seconds
  The total time is measured from the removal of the face mask until bilateral chest rise with the first capnogram upstroke.
Success rate in first attempt | During induction of anesthesia, an average of 60 seconds
  Successful insertion of laryngeal mask airway in a first attempt
Overall success rate | During induction of anesthesia, an average of 60 seconds
  Successful insertion of laryngeal mask airway in a maximum of three attempts
The ease of insertion of device | During induction of anesthesia, an average of 60 seconds
  The ease of placement was assessed using a subjective scale of 1-4 (1= no resistance, 2 = moderate resistance, 3 = high resistance, 4 = inability to place the device)
The number of attempts at insertion of device | During induction of anesthesia, an average of 60 seconds
  The number of attempts for successful insertion of laryngeal mask airway
The ease of gastric tube placement | During induction of anesthesia, an average of 5 minutes
  The ease of gastric tube placement was graded on a subjective scale (1 = easy, 2 = difficult, 3 = unable to pass)
The time for successful gastric tube placement | During induction of anesthesia, an average of 5 minutes
  The insertion time is measured from first handling of the gastric tube to confirmation of its position in the stomach by aspiration of gastric fluid.
The grade of fiberoptic bronchoscopic view | During induction of anesthesia, an average of 5 minutes
  The fiberoptic bronchoscopic view is defined as Grade 1, larynx only seen; Grade 2, larynx and epiglottis posterior surface seen; Grade 3, larynx, and epiglottis tip or anterior surface seen-visual obstruction of epiglottis to larynx: < 50%; Grade 4, epiglottis down-folded, and its anterior surface seen-visual obstruction of epiglottis to larynx: > 50%; Grade 5, epiglottis downfolded and larynx cannot be seen directly.
Peak inspiratory pressure | At 5 minute after insertion of laryngeal mask airway
  Peak inspiratory pressure is recorded from mechanical ventilator.
The number of airway maneuvers required to maintain airway patency | During the surgery, an average of 2 hours after anesthesia induction
  Airway maneuvers required to maintain airway patency, including jaw thrust, head/neck extension and/or device adjustments such as advancement/withdrawal of device, and alterations to cuff volume.
The type of airway maneuvers required to maintain airway patency | During the surgery, an average of 2 hours after anesthesia induction
  Airway maneuvers required to maintain airway patency, including jaw thrust, head/neck extension and/or device adjustments such as advancement/withdrawal of device, and alterations to cuff volume.
Intraoperative complications | During the surgery, an average of 2 hours after anesthesia induction
  Intraoperative complications including coughing, laryngospasm, bronchospasm, hypoxia (SpO2 < 90%), regurgitation, aspiration, blood staining of the device.
Postoperative complications | An average of 2 hours after extubation
  Postoperative complications including sore throat, hoarseness/dysphonia, jaw, neck or ear pain, persistent cough, tachypnea, stridor, hypoxia (SpO2 < 90%), nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyong Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided